CLINICAL TRIAL: NCT03280602
Title: Randomzied Controlled Trial Comparing Tension Band Wiring and Plate Fixation in the Treatment of Olecranon Fractures in Adults
Brief Title: Operative Treatment of Olecranon Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kaare Sourin Midtgaard, Consultant orthopedic surgeon, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/671
Record Dates: First submitted 2017-09-09; First posted 2017-09-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Olecranon Fracture
MeSH Terms: conditions — Olecranon Fracture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Semi-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tension band wiring (TBW) (Active Comparator): TBW following the AO principles with 2 x 1.6 mm K-wires and wire wire cerclage.
  Interventions: Procedure: Tension band wiring (TBW); Procedure: Plate fixation
- Plate fixation (Active Comparator): Plate fixation with Syntes VA-LCP olecranon plates 2.7/3.5
  Interventions: Procedure: Tension band wiring (TBW); Procedure: Plate fixation

INTERVENTIONS:
Procedure: Tension band wiring (TBW) — 2 x K-wire fixation (1.6 mm) and wire cerclage.
Procedure: Plate fixation — Olecranon fractures in this arm are fixed with Synthes´ VA-LCP Olecranon Plates 2.7/3.5.

SUMMARY:
The incidence of olecranon fractures is 12 per 100.000. Traditionally, isolated olecranon fractures have been treated with tension band wiring (TBW). There is a trend towards increased use of plate fixation, though TBW has yielded good and comparable patient reported outcomes. The latter method is substantially cost-effective, but higher complication reports have been reported. There are only two randomized controlled trials comparing TBW and plate fixation, and the literature is inconclusive in which fixation method is preferable in the treatment of olecranon fractures. In this multi-center trial, adult patients (18-75 years) with isolated olecranon fractures will be randomized to either TBW or plate fixation.

DETAILED DESCRIPTION:
Introduction:

The incidence of proximal ulna fractures is 12 per 100.000, and 10 % of all fractures in the upper extremity involve the olecranon. There are several systems classifying olecranon fractures. One of the most frequently used is the Mayo classification system as described by Cabanela and Morrey. Tension band wiring (TBW) is the most common operative technique for the treatment of olecranon fractures, and is said to be the gold standard in the treatment of non-comminuted and minimally comminuted displaced olecranon fractures. Treatment with TBW has shown good clinical results, but due to the thin layer of tissue overlying the proximal ulna, hardware issues are common. The frequency of hardware removal following TBW has been reported as high as 82 %. Only two randomized trials have compared TBW and plate fixation of olecranon fractures. Hume and Wiss compared TBW with one-third tubular plate fixation. The authors found no significant functional differences between the treatment methods, but the rate of symptomatic hardware problems was higher in the group treated with TBW. The authors also noted that loss of reduction was higher in the TBW group at final follow-up (12 months after surgery). Duckworth found no difference in patient reported outcome after one year. The sophistication in plate fixation has evolved since Hume and Wiss published their 25 years ago. The use of locking stable plate fixation in the treatment of olecranon fractures is preferred by many surgeons, especially when treating osteoporotic individuals and in cases with severe fracture fragmentation. Though locking stable implants have shown to improve fragment fixation in biomechanical and cadaveric studies, better patient reported outcome in clinical studies has yet to be proven. It is still unclear if all comminuted fractures should be treated with plate fixation, or if moderately comminuted fractures can be treated with TBW. Hardware related issues following plate fixation have also been described as a frequent problem, and rates of hardware removal up to 56 % have been reported. When approaching the issue of symptomatic hardware problems following TBW and plate fixation, one must take into consideration that the magnitude of secondary surgery is different. The removal of the two K-wires is less extensive than removing an angular stable plate fixation. Removal of symptomatic pin protrusion can be achieved in local anesthesia at the outpatient clinic, whereas plate removal routinely is done in the operating theatre, and usually requires that patient is in regional or general anesthesia. Of course, if the wire cerclage has to be removed in addition to the K-wires, the scope of the procedure is more comparable. There are strong indications that locking plate fixation yield better results when treating severely comminuted olecranon fractures, but the investigators do not know if these modern implants are superior in the treatment of moderately comminuted fractures. Even so, there is a trend toward treating all comminuted olecranon fractures with plate fixation, but the clinical evidence supporting this is limited. The investigators believe there is a need for a robust investigation in the treatment of olecranon fractures to identify the fracture patterns that adequately can be treated with TBW and the ones that should be treated with locking plate fixation.

Study aims:

The investigators want to compare an angular stable plate fixation with TBW in a randomized, controlled multi-center trial. Our hypothesis is that TBW is non-inferior in the treatment of Mayo type IIA and IIB fractures compared with an angular stable implant. The primary outcome measure is the Quick Disability of the Arm, Shoulder and Hand outcome measure (QuickDASH) at 12 months

Study design and methodology:

The study is a randomized, controlled, multicenter trial. Adult patients (18-75 years) admitted with a displaced olecranon fracture in need of surgery will be randomized to either TBW or plate fixation. The design is semi-blinded. At follow-up, an independent investigator will perform an interview and blinded functional examination, followed by an un-blinded examination and interview. Patients will be recruited at the Oslo University Hospital, and other hospitals in the region has been invited to participate in the trial. An experienced trauma surgeon will verify that the fracture meets the inclusion criteria, and the patient will be given thorough oral and written information. After signed consent, the randomization allocation to treatment method will be performed by means of a web-solution made by NTNU WebCRF system with the approval from the OUS Head of Patient Security. To secure an even dispersion in regard to age of the patients and fracture pattern, the inclusion of study patients will be stratified. This will achieve an equal randomization dispersion of patients in in the age interval from 18 to 50 years, and 50 to 75 years. Comminuted and non-comminuted fracture fractures will be randomized in the same fashion.

Power analysis and sample size:

Using the mean value of QuickDASH following olecranon fracture in a similar population, the investigators found the standard deviation (SD) to equal 12 points. The minimal clinical important difference (MCID) has been set to 8 points, and the non-inferiority limit is DASH reduction of 10 points. Level of significance (α) equals 0.05. To prove non-inferiority, a power of 0.90 and with non-inferiority limit at 10, the number required in each group is 39 patients. Taking into account a predicted loss of patients during follow-up, the investigators aim to include at least 45 patients in each group.

Follow-up:

The study patients will be followed-up over a one year period (6 weeks, 12 weeks, 12 months). The rate of hardware removal in both groups will be recorded, and the indication for removal (pain, skin protrusion/wound problems, nerve irritation etc.) will be registered and categorized. All other reoperations will be recorded as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 18 and 75 years with an olecranon fracture Mayo type IIA or IIB will be eligible for inclusion.

Exclusion Criteria:

* Patients younger than 18 or older than 75 years of age.
* Unable to receive oral and written information.
* Concomitant fracture in the injured extremity.
* When the olecranon fracture extends distal to the coronoid process.
* Previous injury or illness in the injured upper extremity with permanent reduced elbow function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
The Quick Disability of the Arm, Shoulder and Hand Outcome Measure (QuickDASH) | 12 months
  The QuickDASH questionnaire evaluates difficulty performing specific tasks and symptoms, social and work function, sleep and confidence. Scaling is ranked from 0 indicating least disability to 100 indicating most disability.

SECONDARY OUTCOMES:
Mayo Elbow Performance Score (MEPS) | 12 months
  MEPS is the primary outcome parameter. MEPS consist of four categories evaluating pain, range of motion, stability and function.6 The scale ranges from 0 to 100, with higher score indicating better outcome. Pain is weighed highest of the 4 variables. Patient outcome can be categorized into excellent (MEPS > 90), good (MEPS 75-90), fair (MEPS 60-74) and poor (MEPS < 60).
Grip strength | 12 months
  A hand dynamometer will be used to measure grip strength in both hands
Range of motion (ROM) | 12 months
  A goniometer will be used to register ROM in elbow flexion, extension and rotation.
The EuroQol five dimensions questionnaire (EQ-5D-5L) | 12 months
  Health status is measures health status/quality of life into one of five levels for the five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The data is computed to a number (EQ-Index) ranging from 0-1.00, where 1.00 is the best possible outcome, and negative values describe a status theoretically worse than being dead. In addition, the patients score their overall life quality on a vertical line, directly measured in millimeters as EQ-VAS score (0-100, 100 best).
Satisfaction with elbow function | 12 months
  An individual satisfaction assessment will be recorded using a visual analogue scale (VAS) of elbow function at follow-up. Zero indicating minimal satisfaction, and 100 indicating maximal satisfaction.
Subjective pain on a scale from 0 (no pain) to 100. | 12 months
  An individual pain assessment will be recorded using a visual analogue scale (VAS) of elbow pain at follow-up. Zero indicating no pain, and 100 indicating maximal pain.
Complications | 12 months
  The patient charts will be reviewed for reports of neurological deficiencies, and an examination of neurologic function will be performed at follow-up. Scar problems, infections, non- and mal-unions and hardware issues will also be reviewed and reexamined. The definition of infection is:
  1. Less serious infection: Superficial wound infection with sign of skin inflammation and/or positive bacterial culture, without the need for secondary surgery, i.e. surgical debridement.
  2. Serious infection: Any postoperative wound infection or sign of deep infection that require secondary surgery.
Hardware removal | 12 months
  Rates of planned and performed hardware removal.
Radiographic evaluation | 12 months
  Radiographs and computer tomographic (CT) scan will be obtained pre- and postoperatively for optimal classification. Radiographs will also be obtained at six weeks, 3 months, and 12 months. Plain x-rays will include true antero-posterior and lateral projections. The fracture pattern will be classified according to the Mayo classification and Schatzker classification. All radiographs will be reviewed and classified by two senior orthopedic trauma surgeons. Assessment of union and non-union will be assessed and recorded. Displacement of the fracture fragments is to be registered in millimeters at the level of the joint. The joint congruency following surgery and at the following radiographs will be evaluated. Osteoarthritis will be classified according to the system of Broberg and Morrey. Heterotopic ossification will be classified according to Hastings and Graham.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duckworth AD, Clement ND, White TO, Court-Brown CM, McQueen MM. Plate Versus Tension-Band Wire Fixation for Olecranon Fractures: A Prospective Randomized Trial. J Bone Joint Surg Am. 2017 Aug 2;99(15):1261-1273. doi: 10.2106/JBJS.16.00773. PMID 28763412
- [Background] Hume MC, Wiss DA. Olecranon fractures. A clinical and radiographic comparison of tension band wiring and plate fixation. Clin Orthop Relat Res. 1992 Dec;(285):229-35. PMID 1446443
- [Background] Buijze G, Kloen P. Clinical evaluation of locking compression plate fixation for comminuted olecranon fractures. J Bone Joint Surg Am. 2009 Oct;91(10):2416-20. doi: 10.2106/JBJS.H.01419. PMID 19797577
- [Background] Chalidis BE, Sachinis NC, Samoladas EP, Dimitriou CG, Pournaras JD. Is tension band wiring technique the "gold standard" for the treatment of olecranon fractures? A long term functional outcome study. J Orthop Surg Res. 2008 Feb 22;3:9. doi: 10.1186/1749-799X-3-9. PMID 18294381
- [Background] Duckworth AD, Clement ND, Aitken SA, Court-Brown CM, McQueen MM. The epidemiology of fractures of the proximal ulna. Injury. 2012 Mar;43(3):343-6. doi: 10.1016/j.injury.2011.10.017. Epub 2011 Nov 9. PMID 22077988
- [Background] Baecher N, Edwards S. Olecranon fractures. J Hand Surg Am. 2013 Mar;38(3):593-604. doi: 10.1016/j.jhsa.2012.12.036. PMID 23428192
- [Background] Edwards SG, Martin BD, Fu RH, Gill JM, Nezhad MK, Orr JA, Ferrucci AM, Love JM, Booth R, Singer A, Hsieh AH. Comparison of olecranon plate fixation in osteoporotic bone: do current technologies and designs make a difference? J Orthop Trauma. 2011 May;25(5):306-11. doi: 10.1097/BOT.0b013e3181f22465. PMID 21464739
- [Background] Karlsson MK, Hasserius R, Karlsson C, Besjakov J, Josefsson PO. Fractures of the olecranon: a 15- to 25-year followup of 73 patients. Clin Orthop Relat Res. 2002 Oct;(403):205-12. PMID 12360028
- [Background] Matar HE, Ali AA, Buckley S, Garlick NI, Atkinson HD. Surgical interventions for treating fractures of the olecranon in adults. Cochrane Database Syst Rev. 2014 Nov 26;2014(11):CD010144. doi: 10.1002/14651858.CD010144.pub2. PMID 25426876
- [Background] Rommens PM, Kuchle R, Schneider RU, Reuter M. Olecranon fractures in adults: factors influencing outcome. Injury. 2004 Nov;35(11):1149-57. doi: 10.1016/j.injury.2003.12.002. PMID 15488508
- [Background] Snoddy MC, Lang MF, An TJ, Mitchell PM, Grantham WJ, Hooe BS, Kay HF, Bhatia R, Thakore RV, Evans JM, Obremskey WT, Sethi MK. Olecranon fractures: factors influencing re-operation. Int Orthop. 2014 Aug;38(8):1711-6. doi: 10.1007/s00264-014-2378-y. Epub 2014 Jun 4. PMID 24893946
- [Background] Tarallo L, Mugnai R, Adani R, Capra F, Zambianchi F, Catani F. Simple and comminuted displaced olecranon fractures: a clinical comparison between tension band wiring and plate fixation techniques. Arch Orthop Trauma Surg. 2014 Aug;134(8):1107-14. doi: 10.1007/s00402-014-2021-9. Epub 2014 Jun 17. PMID 24935660
- [Background] Wagner FC, Konstantinidis L, Hohloch N, Hohloch L, Suedkamp NP, Reising K. Biomechanical evaluation of two innovative locking implants for comminuted olecranon fractures under high-cycle loading conditions. Injury. 2015;46(6):985-9. doi: 10.1016/j.injury.2015.02.010. Epub 2015 Feb 18. PMID 25771445
- [Background] Gruszka D, Arand C, Nowak T, Dietz SO, Wagner D, Rommens P. Olecranon tension plating or olecranon tension band wiring? A comparative biomechanical study. Int Orthop. 2015 May;39(5):955-60. doi: 10.1007/s00264-015-2703-0. Epub 2015 Feb 25. PMID 25711396
- [Background] Wilson J, Bajwa A, Kamath V, Rangan A. Biomechanical comparison of interfragmentary compression in transverse fractures of the olecranon. J Bone Joint Surg Br. 2011 Feb;93(2):245-50. doi: 10.1302/0301-620X.93B2.24613. PMID 21282766